CLINICAL TRIAL: NCT05678010
Title: A Phase I Study Assessing the Safety and Tolerability of Ascending Doses of AZD1390 in Combination With Stereotactic Body Radiation Therapy (SBRT) in Patients With Metastatic Solid Tumor Malignancies
Brief Title: A Study of AZD1390 and Stereotactic Body Radiotherapy (SBRT) for People With Metastatic Solid Tumor Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 22-042
Record Dates: First submitted 2022-12-28; First posted 2023-01-10 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Solid Tumor; Metastatic Solid Tumor; Solid Carcinoma; Solid Tumor, Adult; Metastatic Tumor; Metastatic Cancer
Keywords: Solid Tumor; Metastatic Solid Tumor; Solid Carcinoma; Metastatic Tumor; Metastatic Cancer; 22-042; Memorial Sloan Kettering Cancer Center; AZD1390
MeSH Terms: conditions — Neoplasm Metastasis | interventions — AZD1390; Radiosurgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Arm A, Dose Level 1 (Experimental): Participants have peripheral metastases only, without bowel and lung in SBRT treatment planning target. Once 2 dosing cohorts of safety data are available from concomitant dosing of AZD1390 with SBRT in Arm A, and provided that Arm A is advancing to Cohort 3, Arm B (with bowel and lung in SBRT treatment planning target [PTV]) may be triggered at the initial dose level).
  Interventions: Drug: AZD1390; Radiation: Stereotactic Body Radiotherapy
- Arm A, Dose Level 2 (Experimental): Participants have peripheral metastases only, without bowel and lung in SBRT treatment planning target. Once 2 dosing cohorts of safety data are available from concomitant dosing of AZD1390 with SBRT in Arm A, and provided that Arm A is advancing to Cohort 3, Arm B (with bowel and lung in SBRT treatment planning target [PTV]) may be triggered at the initial dose level).
  Interventions: Drug: AZD1390; Radiation: Stereotactic Body Radiotherapy
- Arm A, Dose Level 3 (Experimental): Participants have peripheral metastases only, without bowel and lung in SBRT treatment planning target. Once 2 dosing cohorts of safety data are available from concomitant dosing of AZD1390 with SBRT in Arm A, and provided that Arm A is advancing to Cohort 3, Arm B (with bowel and lung in SBRT treatment planning target [PTV]) may be triggered at the initial dose level).
  Interventions: Drug: AZD1390; Radiation: Stereotactic Body Radiotherapy
- Arm A, Dose Level 4 (Experimental): Participants have peripheral metastases only, without bowel and lung in SBRT treatment planning target. Once 2 dosing cohorts of safety data are available from concomitant dosing of AZD1390 with SBRT in Arm A, and provided that Arm A is advancing to Cohort 3, Arm B (with bowel and lung in SBRT treatment planning target [PTV]) may be triggered at the initial dose level).
  Interventions: Drug: AZD1390; Radiation: Stereotactic Body Radiotherapy
- Arm B, Dose Level 1 (Experimental): Participants have peripheral metastasis with bowel and lung in SBRT treatment planning target
  Interventions: Drug: AZD1390; Radiation: Stereotactic Body Radiotherapy
- Arm B, Dose Level 2 (Experimental): Participants have peripheral metastasis with bowel and lung in SBRT treatment planning target
  Interventions: Drug: AZD1390; Radiation: Stereotactic Body Radiotherapy
- Arm B, Dose Level 3 (Experimental): Participants have peripheral metastasis with bowel and lung in SBRT treatment planning target
  Interventions: Drug: AZD1390; Radiation: Stereotactic Body Radiotherapy
- Arm B, Dose Level 4 (Experimental): Participants have peripheral metastasis with bowel and lung in SBRT treatment planning target
  Interventions: Drug: AZD1390; Radiation: Stereotactic Body Radiotherapy

INTERVENTIONS:
Drug: AZD1390 — Dose level 1: 20 Dose level 2: 40 Dose level 3: 60 Dose level 4: 80
Radiation: Stereotactic Body Radiotherapy — Participants will receive Stereotactic Body Radiotherapy/SBRT to 2 sites of metastatic tumors consecutively. The two treatment sites will be randomized to SBRT to one site and SBRT + AZD1390 to the other site. Both sites will receive 30Gy in 5 fractions.
  Other Names: SBRT

SUMMARY:
The purpose of this study is to find out whether AZD1390 combined with stereotactic body radiation therapy/SBRT is a safe treatment for people with metastatic solid tumor cancer

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent
* Aged at least 18 years.
* Karnofsky Performance Score (KPS) of ≥60.
* Histologically confirmed diagnosis of cancer with clear evidence of metastasis on imaging. Confirmation of metastasis by biopsy is preferred but not required.
* Candidates for SBRT delivered as 6Gy x 5 daily fractions to 2 sites of disease. The radiation plan should meet departmental guidelines. Patients can have more than 2 sites of disease. If patient requires RT to other sites of disease this can be done after completion of DLT period.
* Adequate organ system functions, as outlined below:

  * Absolute neutrophil count (ANC) ≥1.0 x 109/L
  * Platelets ≥75 x 109/L
  * Hemoglobin ≥8 g/dL
  * Total bilirubin ≤1.5 times the ULN
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 times the ULN if no liver involvement or ≤5 times the ULN with liver involvement with metastatic disease.
  * Creatinine <1.5 times ULN concurrent with creatinine clearance >50 mL/min (measured or calculated by Cockcroft and Gault equation); confirmation of creatinine clearance is only required when creatinine is >1.5 times ULN.
  * Lipase within normal limits (WNL)
  * Creatine kinase (CK) ≤5 times ULN
* Females of childbearing potential must have a negative pregnancy test during screening and must not be breastfeeding or intending to become pregnant during the study. Male patients with female partners of child-bearing potential must be willing to use two forms of acceptable contraception, including one barrier method, during their participation in this study and for 16 weeks following the last dose of the study drug.
* Ability to swallow and retain oral medication.

Exclusion Criteria:

* Prior radiotherapy to the same region within the last 3 months.
* Ongoing treatment for brain metastases. Patients with brain metastases may participate in this trial however, treatment for brain metastases will have to be completed prior to study enrollment. Treatments can begin or resume two weeks after completing protocol therapy.
* History of epilectic disorder.
* For Arm B patients with cancers involving the spinal cord, the length of the spinal cord lesion requiring palliative treatment is greater than 10 cm.
* Past medical history of interstitial lung disease (ILD), drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease.
* Evidence of established ILD on screening CT scan.
* Evidence of severe pulmonary infections, as judged by the investigator, based on clinical findings and investigations.
* Concurrent severe and/or uncontrolled medical condition (e.g., severe COPD).
* Cardiac dysfunction defined as: Myocardial infarction within six months of study entry, NYHA Class II/III/IV heart failure, unstable angina or unstable cardiac arrhythmias.
* Any of the following cardiac criteria:

  * Mean resting corrected QT interval (QTcF) > 470 msec obtained from 3 electrocardiograms (ECGs) (QTc interval will be calculated using Fridericia's formula).
  * Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG, e.g., complete left bundle branch block, third degree heart block.
  * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years-of-age. Patients stable on concomitant medications known to prolong the QT interval may be allowed to participate in the study provided that their mean resting corrected QT interval \(QTcF) is < 470 msec at baseline.
* History or presence of myopathy or raised CK >5 x ULN on 2 occasions at screening.
* Anticancer therapy within 7 days of first SBRT. These treatments should also be held for 7 days after last dose of SBRT. Patients who have received an immune checkpoint inhibitor within 28 days of first administration of study therapy will be excluded.
* History of hypersensitivity to AZD1390 and excipients or drugs with a similar chemical structure or class to AZD1390.
* Patients receiving treatment with strong inhibitors or inducers of CYP3A4 within 2 weeks before the first dose of AZD1390.
* Patients who require sensitive substrates of BCRP, OATP1B1, MATE1, MATE2K and P-gp such as prazosin, cimetidine, simvastatin, dofetilide, metformin, dabigatran, digoxin and fexofenadine should be avoided while on study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-05-17 (Actual); Primary Completion 2028-05-17 (Estimated); Study Completion 2028-05-17 (Estimated)

PRIMARY OUTCOMES:
Assess participants for toxicities related to study treatment | 1 year
  The primary objective is to assess the safety and tolerability of concurrent AZD1390 with SBRT for patients with solid tumor metastases with solid tumor metastases. Participant toxicities will be assessed using the CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Higginson, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (All Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - University of Washington (Data Collection AND Data Analysis), Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org